CLINICAL TRIAL: NCT02996695
Title: Safety, Tolerability, Immunogenicity and Protective Efficacy Against Naturally-Transmitted Malaria of Infectious, Cryopreserved Plasmodium Falciparum Sporozoites (PfSPZ Challenge) Administered by Direct Venous Inoculation Under Chloroquine Chemoprophylaxis (PfSPZ-CVac), in Malian Adults: A Randomized, Double Blind, Placebo-Controlled Trial
Brief Title: Safety and Efficacy of Sanaria's PfSPZ-CVac in Malian Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 15-0052; HHSN272201300022I
Record Dates: First submitted 2016-12-15; First posted 2016-12-19 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2017-07-19

CONDITIONS: Plasmodium Falciparum Infection
Keywords: Chloroquine Chemoprophylaxis; Efficacy; Immunogenicity; Malaria; Placebo; Plasmodium falciparum Sporozoites; Safety; Tolerability
MeSH Terms: conditions — Malaria | interventions — Artesunate; Chloroquine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 204,800 PfSPZ of PfSPZ Challenge (Experimental): 204,800 PfSPZ of PfSPZ Challenge every 4 weeks x 3 doses by DVI, n=31
  Interventions: Drug: Artesunate; Drug: Chloroquine; Biological: PfSPZ (NF54) Challenge
- NaCl placebo (Placebo Comparator): NaCl placebo every 4 weeks x 3 doses by DVI, n=31
  Interventions: Drug: Artesunate; Drug: Chloroquine; Biological: PfSPZ (NF54) Challenge; Other: Placebo

INTERVENTIONS:
Drug: Artesunate — Artesunate is a succinic ester of artemether.
Drug: Chloroquine — 4-aminoquinolone, antimalarial agent for oral administration
Biological: PfSPZ (NF54) Challenge — Cryopreserved Plasmodium falciparum (Pf) fully infectious sporozoites (SPZ) that have been developed to be used to infect volunteers in controlled human malaria infection (CHMI) to assess the efficacy of antimalarial drugs and vaccines. The PfSPZ (NF54) Challenge contains a laboratory malaria strain isolated from a Dutch traveler to Africa.
Other: Placebo — Placebo
  Arms: NaCl placebo

SUMMARY:
Single site, double-blinded, randomized, placebo-controlled clinical trial of PfSPZ-CVac safety, tolerability, immunogenicity and efficacy against naturally occurring malaria in malaria-exposed Malian adults. The overall goal of the study is to evaluate if a regimen of PfSPZ-CVac (PfSPZ Challenge under chemoprophylaxis) is safe, well-tolerated, and provides sterile protection against naturally-occurring malaria in malaria-experienced adults. The study population includes 62 healthy, malaria-experienced adults aged 18-45 years, inclusive, residing in Bougoula Hameau and surrounding villages, Mali. The primary objective of this study is to assess the safety and tolerability of PfSPZ Challenge compared to placebo among malaria-experienced adults taking chloroquine prophylaxis (PfSPZ-CVac)

DETAILED DESCRIPTION:
This is a single site, double-blinded, randomized, placebo-controlled clinical trial of PfSPZ-CVac safety, tolerability, immunogenicity and efficacy against naturally occurring malaria in malaria-exposed Malian adults. The overall goal of the study is to evaluate if a regimen of PfSPZ-CVac (PfSPZ Challenge under chemoprophylaxis) is safe, well-tolerated, and provides sterile protection against naturally-occurring malaria in malaria-experienced adults. Participants will receive three immunizing PfSPZ Challenge injections via direct venous inoculation (DVI) four weeks apart under chloroquine chemoprophylaxis. The PfSPZ Challenge dose will be 204,800 PfSPZ. This is based on results of studies in Europe and in Africa. In Tübingen, Germany, 100% of malaria-naïve adults who received three doses of 51,200 PfSPZ every four weeks under chloroquine chemoprophylaxis were protected against homologous controlled human malaria infection (CHMI). At the same time, studies of PfSPZ Vaccine in malaria-experienced adults in Mali and in Tanzania demonstrate that higher doses of PfSPZ are required to demonstrate immunogenicity and high grade protection in malaria-experienced adults that is comparable to that achieved in malaria-naïve adults studied in the USA. For this reason, the dose selected for this study is four-fold higher than the dose used for Tübingen, Germany. Controls will receive 0.9% sodium chloride (NaCl) as placebo. All participants will receive a standard chemoprophylactic regimen of chloroquine (CQ) for 10 weeks. Chloroquine will be given as a loading dose (600mg chloroquine base) two days before the first administration of PfSPZ Challenge, followed by weekly doses of chloroquine (300mg chloroquine base weekly). Participants will also be treated with a 7-day regimen of artesunate (200 mg per day) after the last PfSPZ Challenge dose of 204,800 sporozoites for malaria parasite clearance, one week after the last CQ dose is given. A total of 62 participants will be randomized in a 1:1 ratio to one of two groups and will be inoculated with PfSPZ Challenge or 0.9% NaCl by DVI so that a total of 62 adults will participate in the study. Participants will be recruited from the MRTC's Bougoula-Hameau site. All volunteers recruited will be healthy adults aged between 18 and 45 years. Safety and infectivity data will be collected. Volunteers, clinical and laboratory investigators will be blinded to group allocation. Participants will be followed every four weeks after the last vaccination as outpatients for active malaria diagnosis and treatment. Passive follow-up will be accomplished by continuous availability of study staff onsite to diagnose and treat malaria and other medical issues that arise. The primary objective of this study is to assess the safety and tolerability of PfSPZ Challenge compared to placebo among malaria-experienced adults taking chloroquine prophylaxis (PfSPZ-CVac). The secondary objectives are: 1. to assess the protective efficacy of PfSPZ-CVac against naturally transmitted P. falciparum malaria infection as diagnosed by thick blood smear microscopy, 2. To assess protective efficacy of PfSPZ-CVac against naturally transmitted P. falciparum malaria infection as diagnosed by qPCR, 3. to assess the expanded efficacy of PfSPZ-CVac compared to placebo, and 4. to examine the immune response to P. falciparum malaria infection.

ELIGIBILITY:
Inclusion Criteria:

1. A male or non-pregnant female aged 18-45 years inclusive at the time of screening.
2. For women of childbearing potential, willingness not to become pregnant or breastfeed until one month after the last CQ dose*.

   *Pre-menopausal female participants will be referred to the local family planning clinic, which offers several means of contraception that are approved and recommended by the Mali Ministry of Health. Contraception (male or female condoms, diaphragm or cervical cap with spermicide, intrauterine device, or hormone-based contraceptive) should be started 30 days before the first vaccination and continue until 30 days after last vaccination.
3. Written informed consent obtained from the participant before screening.
4. Available and willing to participate in follow-up for the duration of study.
5. Residing in Bougoula Hameau region and environs.
6. In general good health based on clinical and laboratory investigation.

Exclusion Criteria:

1. Previous vaccination with an investigational malaria vaccine.
2. Use of an investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days before the first study vaccination, or planned use up to 30 days after last vaccination.
3. Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months before the first vaccination*.

   *This includes any dose level of oral steroids, but not inhaled steroids or topical steroids.
4. Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days before the first study vaccination with the exception of tetanus toxoid.
5. Confirmed or suspected immunosuppressive or immunodeficient condition.
6. Confirmed or suspected autoimmune disease.
7. History of allergic reactions or anaphylaxis to chloroquine, 4-aminoquinolone derivatives, artesunate and artemisinin derivatives, vaccinations or to any vaccine component.
8. History of serious allergic reactions to any substance, requiring hospitalization or emergent medical care.
9. History of allergy to any component of the PfSPZ Challenge product, including human serum albumin.
10. Use or planned use of any drug with anti-malarial activity during the course of the study except for antimalarial medication administered by study clinicians.
11. History of splenectomy.
12. Confirmed pregnancy.
13. Laboratory evidence of liver disease (ALT > upper limit of normal).
14. Laboratory evidence of renal disease (serum or plasma creatinine > upper limit of normal).
15. Laboratory evidence of hematologic disease (platelet count <114,000/mm^3 for males and <144,000/mm^3 for females, or hemoglobin <11.2 g/dL for males and <9.5 g/dL for females).
16. Seropositive for hepatitis B surface antigen or hepatitis C virus (hepatitis C antibody).
17. Seropositive for HIV.
18. Sickle cell trait carriage or sickle cell disease.
19. Administration of immunoglobulin and/or any blood products within the three months preceding the first study. vaccination or planned administration during the study period.
20. Simultaneous participation in any other interventional clinical trial.
21. Acute or chronic pulmonary, cardiovascular, hepatic, renal or neurological condition, severe malnutrition, or any other clinical findings that may increase the risk of participating in the study*.

    *As determined by the PI.
22. Has evidence of increased cardiovascular disease risk (defined as > 10 percent, 5 year risk) as determined by the method of Gaziano*.

    *Risk factors include sex, age (years), systolic blood pressure (mm Hg), smoking status, body mass index (BMI, kg/mm^2), reported diabetes status, and blood pressure.
23. Abnormal screening ECG*.

    *Pathologic Q wave and significant ST-T wave changes, left ventricular hypertrophy, non-sinus rhythm except isolated premature atrial or ventricular contractions, right or left bundle branch block, advanced A-V heart block (secondary or tertiary), QT/QTc interval >450 ms.
24. Other condition that in the opinion of the PI would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol.
25. Documented history of non-febrile seizures or atypical (complex) febrile seizures.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2018-06-22 (Actual)

PRIMARY OUTCOMES:
The number of serious adverse events (SAEs) | 45 days
The number of solicited local and systemic adverse events (AE) | Day 12 after vaccination
The number of unsolicited AEs related to study product | Day 12 after vaccination
The severity of solicited local and systemic adverse events (AE) | Day 12 after vaccination
The severity of unsolicited AEs related to study product | Day 12 after vaccination

SECONDARY OUTCOMES:
Antibody titers against P. falciparum circumsporozoite protein (CSP) and other P. falciparum proteins at serology time points | Days 3, 15, 31, 43,59, 71-77,87,245,and 413
Markers of cell-mediated immunity as assessed by cells producing interferon gamma and/or IL-2 | Days 3, 15, 31, 43,59, 71-77,87,245,and 413
Time to P. falciparum parasitemia, detected by qPCR | within six months after the last vaccination
Time to P. falciparum parasitemia, detected by qPCR | within twelve months after the last vaccination
Time to P. falciparum parasitemia, detected by thick blood film microscopy | within twelve months after the last vaccination
Time to P. falciparum parasitemia, detected by thick blood smear microscopy | Within six months after the last vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bamako - Epidemiology of Parasitic Diseases - Malaria Research and Training Center, Sikasso, Mali

REFERENCES:
- [Derived] Coulibaly D, Kone AK, Traore K, Niangaly A, Kouriba B, Arama C, Zeguime A, Dolo A, Lyke KE, Plowe CV, Abebe Y, Potter GE, Kennedy JK, Galbiati SM, Nomicos E, Deye GA, Richie TL, James ER, Kc N, Sim BKL, Hoffman SL, Doumbo OK, Thera MA, Laurens MB; DMID 15-0052 PfSPZ-CVac Study Team. PfSPZ-CVac malaria vaccine demonstrates safety among malaria-experienced adults: A randomized, controlled phase 1 trial. EClinicalMedicine. 2022 Jul 30;52:101579. doi: 10.1016/j.eclinm.2022.101579. eCollection 2022 Oct. PMID 35928033